CLINICAL TRIAL: NCT00984945
Title: Phase 1 Single Centre, Double-blind, Randomized, Placebo-controlled, Dose-escalation Study of Plant-based H5 VLP (Virus-like Particles), (H5N1) Pandemic Influenza Vaccine Adjuvanted With Aluminium Hydroxide and Administered to Healthy Adults 18-60 Years of Age
Brief Title: Safety Study of a Plant-based H5 Virus-Like Particles (VLP) Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Dr Brian Ward, MUHC Vaccine Study Centre, 14770 Pierrefonds Blvd., Suite 204, Pierrefonds, Quebec, H9H 4Y6
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Medicago H5VLP-001
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-04

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: pandemic vaccine; influenza; H5N1; Virus Like Particle (VLP)
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- H5 VLP vaccine 5 µg (Active Comparator)
  Interventions: Biological: H5 VLP pandemic influenza vaccine 5 µg
- H5 VLP vaccine 10 µg (Active Comparator)
  Interventions: Biological: H5 VLP pandemic influenza vaccine 10 µg
- H5 VLP vaccine 20 µg (Active Comparator)
  Interventions: Biological: H5 VLP pandemic influenza vaccine 20 µg
- Placebo (Formulation buffer) (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H5 VLP pandemic influenza vaccine 5 µg — 0.5 mL, IM, 2 injections 21 days apart
  Arms: H5 VLP vaccine 5 µg
Biological: H5 VLP pandemic influenza vaccine 10 µg — 0.5 mL, IM, 2 injections 21 days apart
  Arms: H5 VLP vaccine 10 µg
Biological: H5 VLP pandemic influenza vaccine 20 µg — 0.5 mL, IM, two injections 21 days apart
  Arms: H5 VLP vaccine 20 µg
Biological: Placebo — 0.5 mL, IM, two injections 21 days apart
  Arms: Placebo (Formulation buffer)

SUMMARY:
The primary objective is to assess the safety and tolerability of two consecutive doses of plant-based H5 VLP, (H5N1) pandemic influenza vaccine combined with Alhydrogel®, given 21 days apart, at three dose levels: 5µg, 10µg and 20µg., compared to the placebo, and combined with Alhydrogel®.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 to 60 years of age
* Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, vital signs, screening laboratories and medical history conducted no more than 30 days prior to study vaccine administration
* BMI of ≥18 and ≤29
* Comprehension of the study requirements, expressed availability for the required study period and ability to attend scheduled visits
* Accessible by telephone on a consistent basis
* In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee
* If female and capable of child-bearing, have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

  1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration
  2. Requiring a change in medication dosage in one month prior to test article administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  3. Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to test article administration
* Any medical or neuropsychiatric condition which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting
* Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection or presence of lymphoproliferative disease
* Presence of any febrile illness, oral temperature of >38.0 C within 24 hours of test article administration. Such subjects may be re-evaluated for enrolment after resolution of illness
* History of autoimmune disease
* Administration of any vaccine (including any other influenza vaccine) within a 30 day period prior to study enrolment, or planned administration within the period from the first vaccination up to blood sampling at Day 42 or within 30 days prior to blood sampling at Day 228. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to test article administration. Receipt of any other emergency immunizations (e.g. rabies) will result in a case-by-case review of continued participation.
* Use of any investigational or non-registered product within 90 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other drug study while participating in this study
* Treatment with systemic glucocorticoids at a dose exceeding ≥ 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of first test article administration, or any other cytotoxic or immunosuppressant drug or any immune globulin preparation within three months of vaccination. Nasal or inhaled glucocorticoids are allowed
* Any significant disorder of coagulation or treatment with coumadin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin, and without a clinically apparent bleeding tendency are eligible
* History of previous H5N1 vaccination
* History of allergy to any of the constituents of H5 VLP (H5N1) study vaccine, Alhydrogel® (aluminium hydroxide), or the phosphate buffer.
* History of severe allergic reactions or anaphylaxis
* History of tobacco allergy
* Have received a blood transfusion or immunoglobulins within 90 days of study entry
* If female, and of childbearing potential, has not been consistently using effective birth control for the 28 days prior to study entry. An example of highly effective birth control is oral contraceptives, hormone implants, abstinence (confirmed by Investigator), or male condom plus spermicide. All female subjects, regardless of birth control history must provide a urine sample for pregnancy screening. Effective birth control must be used for the duration of the study. The subject must have no plan to become pregnant during the study period. Females who are post-menopausal (no spotting at all) for at least two (2) years will not require a urine pregnancy test.
* Among female subjects, either known pregnancy or urine beta-human chorionic gonadotropin (ß-hCG) test results consistent with pregnancy prior to test article administration on Day 0
* Female subjects who are lactating
* Vital sign abnormalities: systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥90 mmHg, resting pulse rate <40 bpm or >100 bpm
* Cancer or treatment for cancer within 3 years of test article administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated through reported adverse events, physical examination findings; clinical laboratory results and vital signs. | 21 days

SECONDARY OUTCOMES:
The secondary objective is to evaluate the immunogenicity of two consecutive doses of plant-based H5 VLP vaccine combined with Alhydrogel®, at three dose levels: 5µg, 10µg and 20µg, compared to the placebo, combined with Alhydrogel®. | 21days after each vaccination and 6-month after boost injection

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ward, MD, Principal Investigator — MUHC Vaccine Study Centre
Locations (1):
- MUHC Vaccine Study Centre, Pierrefonds, Quebec, Canada

REFERENCES:
- [Derived] Landry N, Ward BJ, Trepanier S, Montomoli E, Dargis M, Lapini G, Vezina LP. Preclinical and clinical development of plant-made virus-like particle vaccine against avian H5N1 influenza. PLoS One. 2010 Dec 22;5(12):e15559. doi: 10.1371/journal.pone.0015559. PMID 21203523